CLINICAL TRIAL: NCT02375945
Title: Prospective, Randomized Controlled Trial Comparing the Effect of a Non-elastic Compression Device Juxta Reduction Kit (Medi ®)" Versus Elastic Class 1 Stockings (BSN Medical® in Patients Undergoing Total Knee Arthroplasty
Brief Title: Comparison Between a Non-elastic Falcro Device and Current Method After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, principal investigator, Nij Smellinghe Hosptial
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NS7NL
Record Dates: First submitted 2015-02-07; First posted 2015-03-03 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Lymphedema
Keywords: lymphedema; post operative compression treatment; compression therapy; adjustable fulcro wraps; edema
MeSH Terms: conditions — Lymphedema; Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- current compression stocking Comprinet® (Active Comparator): Immediately post operatively 24 hours compression therapy starts with "Elastomull Haft ®", an elastic bandage, combined with a Comprinet stocking (BSM Medical®) for anti thrombotic purposes. The anti thrombosis stocking is worn 6 weeks post operatively. After 4 hours the patient is ambulated and the physical therapy starts.
  Interventions: Device: New non-elastic compression kit; Device: current compression stocking Comprinet®
- New non-elastic compression kit (Experimental): Juxta Reduction Kit ® Immediately post operative compression starts with the Juxta Reduction Kit® for the knee region, combined with an anti thrombosis stocking (Struva 2, for prevention of trombo-embolism). Both the stocking and the Juxtra Pro are used for six weeks. After 4 hours the patient ambulated and the physical therapy starts.
  For the first 24 hours and longer if necessary (depending on the skills of the patient) Juxta experienced staff will apply the device and the fit and the use of the device will be checked.
  In the second phase between approximately 24 hours and 6 weeks patients may adjust the Juxta-pro according to their needs and comfort by themselves.
  Interventions: Device: New non-elastic compression kit; Device: current compression stocking Comprinet®

INTERVENTIONS:
Device: New non-elastic compression kit — Comparison of new non-elastic bandage kit with the currently accepted method
  Other Names: study material
Device: current compression stocking Comprinet® — Comparison of new non-elastic bandage kit with the currently accepted method

SUMMARY:
Swelling is a common problem after knee arthroplasty often leading to delayed wound healing, lasting functional impairment and hematoma.

Due to this complications, sometimes the risk for deep venous thrombosis is raised. This study investigates a new self adjustable device to reduce swelling more effective postoperatively. The investigators compare the new device to the current general practice by using a standard class 1 elastic stocking

DETAILED DESCRIPTION:
Purpose Pain, swelling and inflammation are expected during early recovery from total knee arthroplasty (TKA). Compression therapy is a frequently used modality in the direct post operative treatment, but there is a great variety in the use of materials, the way and time frame of application. The most common goals of the compression therapy are prevention and reduction of the swelling. At the same time the literature is not consistent about the use and effects of compression therapy other than for prevention of trombo-embolic processes The state of the art care concepts for patients undergoing a total knee arthroplasty embraces the concept of "fast track" (Kehlet et al) with important parts as early mobilisation and optimal analgesics. In the investigators hospital this concept has already been implemented.

During the stay in the hospital the challenge is to give adequate compression therapy to prevent and reduce swelling and enhance woundhealing. At the same time it is essential to optimise ambulation of the patient and the possibilities to exercise.

The current protocol in the investigators hospital consists of 24 hours compression therapy with "Elastomull Haft ®", an elastic bandage for the knee region, combined with a Comprinet stocking (BSM Medical®) for anti thrombotic purposis. The anti thrombosis stocking is worn for a period of 6 weeks.

The compression is combined with the use of the Continious Passive Motion device for 4 hours post operatively (2 hours immobilisation in a position of 90 degrees flexion, followed by 2 hours hours of passive motion in a range of 60-90 degrees flexion). Four hours post operatively the patient is ambulatend and the physical therapy starts.

The investigators wonder if this is the optimal way of post-operative care. Swelling of the knee and the whole leg can remain a problem in the first 6 weeks of recovery which inhibits rehabilitation. Sometimes delayed woundhealing will occur and patients may complain of more durable pain which make analgesics necessary.

Prolonging adequate compression could improve the post-operative course and support the total rehabilitation process.

The "Juxta Reduction Kit (by Medi) ®" , applied for the knee could be an adequate solution to replace the current protocol of compression therapy.

The "Juxta Reduction Kit ®" is a non-elastic compression device which can be tailored (by cutting it to the correct size) to the circumference of the leg prior to the operation. Direct post operatively the compression device can be adjusted by the staff and in the following days patients are enabled to adjust the device by themselves by using the Velcro ties to loosen or fasten it.

The device is suitable in early mobilisation and gives the patient tools for selfmanagement of the compression by using the Velcro flaps. The material doesn't restrict the range of motion and so the possibility to ambulate and to exercise as advised in the fast track concept is optimised.

In this study the patients will use the compression device for a period of six weeks in combination with an anti thrombosis stocking (Struva class 2) Outcome parameters will be measured in a scheduled way, described in scheme 1.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing a primary elective total knee arthroplasty
* The patient is able to understand the study and is willing to give written informed consent to the study.

Exclusion Criteria:

* Allergy against one of the used materials
* Severe systemic diseases causing peripheral oedema
* Acute superficial or deep vein thrombosis
* Arterial occlusive disease (stadium II, III or IV) ABPI<0,8
* Local infection in the therapy area
* auto-immunological disorders or vasculitis
* use of systemic corticosteroids
* Inability to don, doff, and adjust the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
efficacy of the device on wound healing, swelling reduction and functional improvement | 12 weeks
  efficacy of the device on wound healing, swelling reduction and functional improvement
circumference measurements | 12 weeks
  efficacy of the device

SECONDARY OUTCOMES:
comfort to the patient / QoL | 12 weeks
  The effects and wearing comfort to the patient is closely recorded. Further the number of adjustment of the device by the patient and his/her experience

CONTACTS AND LOCATIONS:
Locations (1):
- Nij Smellinghe hospital, Drachten, Provincie Friesland, Netherlands